CLINICAL TRIAL: NCT00961142
Title: Multicenter Phase II Study of Haploidentical Hematopoietic Cell Transplantation With CD3/CD19 Depleted Grafts After a Reduced Intensity Conditioning Regimen for Adult Patients With Acute Leukemia
Brief Title: Haploidentical Stem Cell Transplantation With CD3/CD19 Depletion and Reduced Intensity Conditioning in Patients With Acute Leukemia
Acronym: CD3/CD19 Haplo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Wolfgang Bethge, Prof. Dr., University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2007-006016-33
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Haploidentical Transplantation; CD3/CD19 Depletion; AML; ALL; Reduced Intensity Conditioning
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Thiotepa; Melphalan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fludarabine, Thiotepa, Melphalan, Thymoglobuline (ATG) — Conditioning with Fludarabine 30 mg/m2/24h day-8 to -4, Thiotepa 2x5 mg/kg day -3, Melphalan 60 mg/m2 day -2 to -1 and Thymoglobuline (ATG)1.5mg/kg/day day -9 to -6. PBSC depleted of CD3 and CD19 cells by immunomagnetic depletion on CliniMACS.

SUMMARY:
Feasibility and toxicity of haploidentical allogeneic HCT after a reduced intensity conditioning regimen with CD3/CD19 depleted grafts. This study enrolls patients with acute leukemia in complete remission with an indication for allogeneic HCT but without a suitable HLA-identical donor

ELIGIBILITY:
Inclusion Criteria:

* Patients with either ALL or AML in CR with an indication for allogeneic HCT according to the following criteria:
* AML: high risk patients with one or more of the following risk factors:

  * FLT-3 mutation
  * Complex cytogenetics
  * abn(3q), -5/5q-, -7/7q-, abn(12p), abn(17p)
  * Late CR > induction I
  * Age >60
  * Patients in 2.CR
  * Secondary AML
  * Relapse after a preceding allogeneic HCT from an HLA-identical donor
* ALL: high risk patients with one or more of the following risk factors:

  * Pro-B-ALL
  * Initial WBC >30.000/µL
  * CR after day 46 after Induction II
  * Complex cytogenetics, t(9,22), t(4,11)
  * Early or mature T-ALL
  * Initially refractory patients with late CR
  * Rising MRD level
  * Patients in 2. CR
  * Relapse after a preceding allogeneic HCT from an HLA-identical donor
  * No HLA-identical donor (not more than 1 antigen mismatch (9/10-Match) or more than 2 allelic mismatches by high-resolution typing). Critical cases should be discussed with the PI.
  * Age <=65, >=18 years
  * Karnofsky Index >60%

Exclusion Criteria:

* Patients with >5% blasts in BM at the time of transplantation
* Less than 3 months after preceding HCT
* CNS involvement with disease
* History of neurologic impairment such as: seizures, severe peripheral neuropathy, signs of leukoencephalopathy, CNS infection, multiple intrathecal chemotherapies, CNS irradiation. In case of heavy pretreatment with irradiation or intrathecal chemotherapy pretransplant CNS MRI and neurological consultation are mandatory
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month.
* Liver function abnormalities with bilirubin >2 mg/dL and elevation of transaminases higher 2x upper limit of normal.
* Chronic active viral hepatitis
* Ejection fraction <40 % on echocardiography
* Patients with > grade II hypertension by CTC criteria
* Creatinine clearance <50 ml/min
* Respiratory failure necessitating supplemental oxygen or DLCO <30%
* Allergy against murine antibodies
* HIV-Infection
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control during study treatment and for at least 12 months thereafter. (Women of childbearing potential must have a negative serum pregnancy test at study entry)
* Concurrent severe and/or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study
* Patients with a history of psychiatric illness or condition which could interfere with their ability to understand the requirements of the study (this includes alcoholism/drug addiction)
* Patients unwilling or unable to comply with the protocol
* Unable to give informed consent
* Enrollment in an other trial interfering with the endpoints of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment related mortality after haploidentical HCT | 1 year after HCT
  Cumulative Incidence of treatment related mortality

SECONDARY OUTCOMES:
overall survival | 1, 2 and 5 years after inclusion
  by Kaplan-Meier
Evaluate Engraftment | One year after HCT
Evaluate Toxicity | One year after HCT
Evaluate Disease Free Survival | 1, 2 and 5 years after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A. Bethge, MD, Principal Investigator — Medical Center University Hospital Tuebingen
Locations (8):
- Germany (8):
  - University of Dresden Medical Center, Dresden
  - Center for Marrow Transplantation, University of Essen, Essen
  - Medical Center University of Halle, Halle
  - Medical Center University of Hamburg, Hamburg
  - Medical Center University of Muenster, Münster
  - South West German Cancer Center, University of Tuebingen Medical Center, Tübingen
  - Deutsche Klinik für Diagnostik, Wiesbaden
  - University of Wuerzburg Medical Center, Würzburg

REFERENCES:
- [Background] Bethge WA, Faul C, Bornhauser M, Stuhler G, Beelen DW, Lang P, Stelljes M, Vogel W, Hagele M, Handgretinger R, Kanz L. Haploidentical allogeneic hematopoietic cell transplantation in adults using CD3/CD19 depletion and reduced intensity conditioning: an update. Blood Cells Mol Dis. 2008 Jan-Feb;40(1):13-9. doi: 10.1016/j.bcmd.2007.07.001. Epub 2007 Sep 14. PMID 17869547
- [Background] Bethge WA, Haegele M, Faul C, Lang P, Schumm M, Bornhauser M, Handgretinger R, Kanz L. Haploidentical allogeneic hematopoietic cell transplantation in adults with reduced-intensity conditioning and CD3/CD19 depletion: fast engraftment and low toxicity. Exp Hematol. 2006 Dec;34(12):1746-52. doi: 10.1016/j.exphem.2006.08.009. PMID 17157172
- See also: Homepage BMT-Study Group Tuebingen — http://www.onkologie-tuebingen.de/ifa0.htm
- Available data/document: Results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2007-006016-33